CLINICAL TRIAL: NCT03058393
Title: Effectiveness of Teach-back in Orthopedic Treatment Decision Discussions
Brief Title: Analyzing Challenging Clinical Discussions in Orthopaedics
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Extenuating circumstances
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00079809
Record Dates: First submitted 2017-02-14; First posted 2017-02-20 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2018-06

CONDITIONS: Teach-Back Communication; Arthritis; Knee Osteoarthritis; Knee Arthropathy
MeSH Terms: conditions — Teach-Back Communication; Arthritis; Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Teach-Back Group (Experimental): A teach-back lesson will be provided to physician participants (Teach-Back Group), who are participating in challenging clinical discussions with patients
  Interventions: Other: Teach-Back Lesson

INTERVENTIONS:
Other: Teach-Back Lesson — A teach-back lesson will be given to providers (teach-back group) who have challenging clinical discussions with patients

SUMMARY:
The goal of this study is to analyze patient:provider communication surrounding the discussion of difficult clinical conversations such as knee replacement options. This study will also examine how using the teach-back communication technique can improve communication between patients and providers. Orthopedic residents, fellows, physician assistants, and attendings that agree to participate will be consented. Patients, who are likely to engage in a difficult clinical conversation, such as those who have a clinical indication for a Total Knee Replacement or a Partial Knee Replacement, will be recruited from participating providers clinical schedules. Patient:provider interactions will be recorded and then the providers will attend a 1 hour education lecture about how to use teach-back. After attending the lecture, additional patient:provider interactions will be recorded and analyzed via a qualitative approach. Additionally, providers will participate in a semi-structured interview to capture their perceptions of teach-back and what challenges and benefits they may derive from using it.

ELIGIBILITY:
Inclusion Criteria (Patient Participants):

* Age 18 years and older
* Clinical indication for multiple treatment options

Exclusion Criteria (Patient Participants):

* Non-English speaking
* Minors or non-consenting other individuals (spouses, friends, family members, children) in the patient room during the clinical visit

Inclusion Criteria (Provider Participants)

* Age 18 years and older
* A resident, fellow, physician assistant, or attending in the Duke Department of Orthopaedic Surgery

Exclusion criterion (Provider Participants):

• Non-English speaking

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-04-17 (Actual); Primary Completion 2018-11-07 (Actual); Study Completion 2018-11-07 (Actual)

PRIMARY OUTCOMES:
Provider's uninterrupted utterances | End of discussion with patient, 20 minutes
  We will assess this outcome directly from audio-recorded conversations. A coding scheme will then be developed that captures the average length of provider utterance without asking a question or an interruption from a patient
Patient/provider talking ratio | End of discussion with patient, 20 minutes
  This outcome will also be assessed from audio-recorded conversations. The transcript will be coded and the coding scheme will compare how often and how long patients talk compared to provider talking.

SECONDARY OUTCOMES:
Providers perceptions about teach-back | End of semi-structured interview, one hour
  This outcome will be assessed via semi-structured interviews.
Providers belief of future use of teach-back | End of semi-structured interview, one hour
  This outcome will be assessed via the semi-structured interview

CONTACTS AND LOCATIONS:
Overall Officials: Richard C Mather III, MD, MBA, Principal Investigator — Duke University
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No